CLINICAL TRIAL: NCT01486914
Title: A Single Centre, Randomized, Balanced Double Blind, Cross-Over Trial Investigating the Bioequivalence of NovoRapid® Produced by the Current Process and Insulin Aspart With the Same Formulation as NovoRapid®, Produced by the NN2000 Process
Brief Title: Comparison of Insulin Aspart Produced by Current Process and the NN2000 Process
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2000-1512
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NN2000 (Experimental)
  Interventions: Drug: insulin aspart
- IAsp (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Single dose of each formulation administrated subcutaneously (s.c., under the skin) at two separate dosing visits

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare insulin aspart produced by current process and the NN2000 process.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Caucasian
* Normal findings in medical history and physical examination unless the investigator considers any abnormality to be clinically irrelevant
* Fasting blood glucose below or equal to 6 mmol/L
* Body mass index (BMI) 22.0-27.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Participated in another clinical study with an investigational drug within the last 4 weeks
* Any condition requiring the regular use of any medication, including herbal remedies, over the counter medicines and vitamins. Occasional paracetamol is acceptable
* Known or suspected allergy to the trial product or related products
* Family history of type 2 diabetes

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2003-01-19 (Actual); Primary Completion 2003-02-24 (Actual); Study Completion 2003-02-24 (Actual)

PRIMARY OUTCOMES:
Area under the Curve (AUC) (insulin aspart)

SECONDARY OUTCOMES:
Cmax (maximum plasma concentration)
Terminal half life (t½)
Incident of hypoglycaemic episodes
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Manchester, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com